CLINICAL TRIAL: NCT06504732
Title: A Phase II/III Clinical Study Evaluating IAH0968 in Combination or Not in Combination With the CAPEOX Regimen in HER2-expressing Advanced/Metastatic Solid Tumors and Gastric Cancer
Brief Title: To Evaluate IAH0968 in Combination With CAPEOX in HER2-positive Gastric Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: SUNHO（China）BioPharmaceutical CO., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAH0968-203
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-07

CONDITIONS: Stomach Neoplasms; Solid Tumor
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): 10-20 subjects with HER2-positive advanced/metastatic gastric cancer (including adenocarcinoma of the gastro-esophageal junction) without systemic treatment will be enrolled in combination with the CAPEOX regimen at a dose of 15 mg/kg of IAH0968 to assess the safety and tolerability of the combination therapy.
  Interventions: Drug: IAH0968
- Cohort 2 (Experimental): 10-30 subjects with advanced/metastatic malignant solid tumors with low HER2 expression who have failed standard therapy or have no standard therapy will be enrolled at the 20 mg/kg IAH0968 dose to assess the safety and tolerability of IAH0968 monotherapy. The safety of IAH0968 at 15 mg/kg in combination with the CAPEOX regimen will be evaluated if the starting dose group, i.e., exceeds the MTD.
  Interventions: Drug: IAH0968
- Cohort 3 (Experimental): The CAPEOX regimen will be combined at the 20 mg/kg IAH0968 dose to enroll 20-40 unsystematically treated subjects with advanced/metastatic colorectal or gastric cancers with low expression of HER2, including adenocarcinomas of the gastro-esophageal junction, in order to assess the safety and tolerance of the combination therapy. The safety of IAH0968 at 15 mg/kg in combination with the CAPEOX regimen will be evaluated if the starting dose group, i.e., exceeds the MTD.
  Interventions: Drug: IAH0968

INTERVENTIONS:
Drug: IAH0968 — Subjects were treated with IAH0968 in combination with or without the CAPEOX regimen in the corresponding groups. Every 3 weeks was defined as a treatment cycle and IAH0968 was used for a maximum of 35 cycles.

SUMMARY:
The safety, tolerability, and determination of the maximum tolerated dose (MTD) of the combination therapy were first evaluated for IAH0968 in combination with or without the CAPEOX regimen in unsystematically treated subjects with HER2-expressing advanced/metastatic colorectal or gastric cancers (including adenocarcinomas of the gastro-esophageal junction) or HER2-hypo-expressing advanced/metastatic solid tumors. The efficacy of IAH0968 in combination with the CAPEOX regimen versus trastuzumab in combination with the CAPEOX regimen in subjects with HER2-positive advanced/metastatic gastric cancer, including gastro-esophageal junction adenocarcinoma, was then assessed by progression-free survival (PFS) according to the Research and Evaluation Criteria for the Evaluation of Efficacy in Solid Tumors (RECIST) 1.1.

DETAILED DESCRIPTION:
This clinical study is a randomized, multicenter Phase II/III clinical study to investigate the efficacy of IAH0968 in combination or not in combination with the CAPEOX regimen in the treatment of subjects with HER2-expressing advanced/metastatic solid tumors and gastric cancer. The study is divided into two study phases: a Phase II clinical study and a Phase III clinical study.

Adverse events and adverse reactions were assessed in the study through clinical observation, vital signs monitoring, laboratory tests, etc., while PK, ADA and other relevant samples were collected; and using RECIST 1.1 as the standard for tumor assessment, subjects were assessed for tumors every 6 weeks starting from the first infusion of the study drug until the occurrence of disease progression, the initiation of new antitumor therapy, and the judgement of the investigator that it was not suitable for continued participation (e.g., development of intolerable adverse reactions), loss to visit, voluntary withdrawal, death, or study termination/suspension.

Upon withdrawal or termination of treatment (+7 days), subjects should be visited for termination of treatment (except in the case of death and loss to follow-up), as far as possible, prior to the initiation of new antitumor therapy, with relevant laboratory investigations and ADA samples, and thereafter followed up by telephone every 12 weeks (±7 days) for survival (OS) until loss to follow-up or death.

The phase II study was an open-label, nonrandomized clinical study, which was planned to be divided into 3 cohorts.The phase III study used a randomized, parallel-controlled, multicenter study design.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 18~75 years old (including critical mass), gender is not limited. 2) Phase II cohort 1 and III only: patients with locally advanced or metastatic gastric cancer (including adenocarcinoma of the gastro-esophageal junction) diagnosed by histopathology, unsuitable for radical surgical resection or localized treatment, and who have not received systemic antitumor therapy (including systemic chemotherapy, molecularly-targeted drug therapy, biologic therapy, and other investigational therapeutic agents) for GC (except for adjuvant chemotherapy for >6 months), and who have demonstrated disease progression; and patients who have been diagnosed by immunohistochemistry (IHC) staining and/or fluorescence in situ hybridization (FISH). and demonstrated disease progression excepted); HER2 positivity (IHC 3+, or IHC 2+ and FISH +) demonstrated by immunohistochemical (IHC) staining and/or fluorescence in situ hybridization (FISH).

  3) Phase II Cohort 2 only: Have histologically or cytologically confirmed advanced malignant solid tumors that have failed standard treatment, or for which no standard treatment options are available, or for which standard treatment is not applicable at this stage; and are HER2 underexpressed (IHC 2+ and FISH-, or IHC 1+) as evidenced by immunohistochemistry (IHC) staining and/or fluorescence in situ hybridization (FISH).

  4) Phase II Cohort 3 only: with locally advanced or metastatic gastric cancer (including gastro-oesophageal junction adenocarcinoma) or colorectal cancer diagnosed by histopathology, unsuitable for radical surgical resection or localized treatment, with no prior systemic (including systemic chemotherapy, molecularly-targeted drug therapy, biologic therapy, and other investigational therapeutic agents) antitumor therapy (having received adjuvant chemotherapy for >6 months with evidence of disease progression), patients with wild-type KRAS, NRAS, and BRAF genes (mCRC only); and HER2 low expression (IHC 2+ and FISH-, or IHC 1+) demonstrated by immunohistochemical (IHC) staining and/or fluorescence in situ hybridization (FISH).

  5) At least 1 measurable lesion according to RECIST 1.1 criteria (tumor lesions located in the area of prior radiotherapy or other localized regional treatment sites are generally not considered measurable lesions unless the lesion shows definite progression or persists after three months of radiotherapy).

  6) Eastern Cooperative Oncology Group (ECOG) physical status score of 0 to 1. 7) Have an expected survival of ≥ 3 months. 8) Adequate organ function:
  * Hematologic system (no transfusion or hematopoietic stimulating factor therapy within 14 days): absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 90 × 109/L, hemoglobin (HGB) ≥ 90 g/L; Liver function: total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN), except Gilbert's syndrome; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 times the ULN, liver metastasis or hepatocellular carcinoma patients need to AST and ALT ≤ 5.0 times the ULN and total bilirubin ≤ 3.0 times the ULN; Renal function: serum creatinine (Cr) ≤1.5 times ULN; if creatinine >1.5 times ULN, creatinine clearance (Ccr) ≥50 mL/min (calculated according to Cockcroft-Gault formula);

    ④ Coagulation function: International Normalized Ratio (INR) ≤ 1.5 times ULN for prothrombinogen, Activated Partial Thromboplastin Time (APTT) ≤ 1.5 times ULN, or INR and APTT ≤ 2.5 times ULN for patients with liver metastasis or hepatocellular carcinoma.

    9) Eligible patients (male and female) of childbearing potential must agree to use a reliable method of contraception (hormonal or barrier method or abstinence) with their partner for the duration of the trial and for at least 6 months after the last dose; female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of study drug.

    10) Subjects must give informed consent for this study prior to the trial and voluntarily sign a written informed consent form.

Exclusion Criteria:

* 1) Phase II Cohort 2 only: received antitumor therapy such as chemotherapy, radiotherapy, biologic therapy, endocrine therapy, immunotherapy, etc. within 4 weeks prior to the first use of study drug, except for the following:

  * Nitrosourea or mitomycin C within 6 weeks prior to first use of study drug;

    ② Oral fluorouracil analogs and small molecule targeted drugs for 2 weeks prior to the first use of the study drug or within 5 half-lives of the drug (whichever is longer);

    ③ Within 2 weeks prior to first use of the study drug for proprietary Chinese medicines with antitumor indications.

    2) Received other unlisted clinical investigational drug or therapy within 4 weeks prior to first use of the study drug.

    3) Adverse effects of prior antineoplastic therapy have not returned to NCI CTCAE 5.0 grade rating of ≤ grade 1 or relevant provisions of the enrollment criteria (except for toxicities judged by the investigator to pose no safety risk, such as alopecia, grade 2 peripheral neurotoxicity, and hypothyroidism stabilized by hormone replacement therapy).

    4) Known hypersensitivity to any antibody-based drug (NCI CTCAE 5.0 grade rating ≥ 3) or hypersensitivity to the study drug and the active ingredient or inactive excipients of the CAPEOX regimen.

    5) Diagnosed defective mismatch repair (dMMR) or high microsatellite instability (MSI-H) solid tumor (except unknown MSI/MMR status).

    6) Major surgical procedure (excluding puncture biopsy), major trauma within 4 weeks prior to first use of study drug, or need for elective surgery during the trial.

    7) Received systemic glucocorticosteroids (prednisone > 10 mg/day or equivalent) within 14 days prior to the first dose of study drug, except for the following: treatment with topical, ocular, intra-articular, intranasal, and inhaled glucocorticosteroids; and short-term prophylactic glucocorticosteroids (e.g., for prevention of allergy to contrast media).

    8) Other immunosuppressive therapy within 28 days or 5 half-lives (whichever is longer) prior to first use of study drug.

    9) Use of immunomodulatory drugs within 14 days prior to first use of study drug.

    10) Use of any live vaccine within 4 weeks prior to the first dose of study drug.

    11) Previous allogeneic hematopoietic stem cell transplantation or organ transplantation.

    12) Parenchymal brain metastases or meningeal metastases with clinical symptoms.

    13) Have an active infection that currently requires intravenous anti-infective therapy.

    14) Have a history of immunodeficiency, including a positive antibody test for human immunodeficiency virus (HIV).

    15) Have active hepatitis B (HBsAg positive and HBV-DNA positive or greater than the upper limit of normal) and active hepatitis C (hepatitis C virus antibody positive and HCV RNA positive or greater than the upper limit of normal).

    16) Have severe and uncontrollable lung disease (severe infectious pneumonia, interstitial lung disease, etc.).

    17) Have a history of severe cardiovascular disease, including but not limited to:
  * Having severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, degree II-III atrioventricular block;

    * Mean QT interval (QTcF) corrected by the Fridericia method > 470 ms;

      ③ Acute coronary syndrome, congestive heart failure, aortic coarctation, stroke, or other grade 3 or higher cardiovascular event within 6 months prior to the first dose;

      ④ Presence of New York Heart Association (NYHA) Cardiac Function Class ≥ Grade II heart failure or left ventricular ejection fraction (LVEF) < 50%, or other structural heart disease judged by the investigator to be of high risk;

      ⑤ Clinically uncontrolled hypertension. 18) Active, or previous autoimmune disease with potential for relapse (e.g., systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except for clinically stable autoimmune thyroid disease, type I diabetes mellitus, vitiligo, cured atopic dermatitis in children, and psoriasis that does not require systemic therapy (within the past 2 years).

      19) Presence of other malignancies within 5 years prior to the start of study dosing, except: malignancies for which cure can be expected with treatment (including, but not limited to, adequately treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated by radical surgery).

      20) Presence of clinically uncontrollable third interstitial fluid that, in the judgment of the Investigator, makes enrollment inappropriate.

      21) Known alcohol or drug dependence. 22) Have a mental disorder or poor compliance. 23) Pregnant or lactating females. 24) In the opinion of the investigator, the subject has a history of other serious systemic disease or is otherwise unsuitable for enrollment in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experienced At Least One Adverse Event (AE) | Up to approximately 48 months
  An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who experienced at least one AE is presented.
Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE) | Up to approximately 48 months
  An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who discontinued study treatment due to an AE is presented.
Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 48 months
  PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 was calculated using the product-limit (Kaplan-Meier) method for censored data.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No